CLINICAL TRIAL: NCT04907461
Title: Laparoscopic Guided vs Ultrasound Guided Transabdominal Plane Block in Minimal Invasive Colorectal Surgery; a Comparison Between Time of Procedure and Efficacy on Pain Relief and Postoperative Opioid Consumption.
Brief Title: Laparoscopic vs Ultrasound Guided TAP Block in Colorectal Surgery. A Randomised Controlled Study.
Acronym: LAPTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LAPTAP Study
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2022-07

CONDITIONS: Laparoscopic Surgical Procedure; Nerve Block

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. The participants are during surgery randomized to either Laparoscopic guided TAP block or Ultrasound guided TAP block.
Who Masked: Participant
Masking Description: Participants are under narcosis during randomisation and intervention. The surgical staff are aware of randomisation and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic guided TAP block (Experimental): The surgeon uses a laparoscopic technique to visualise the peritoneum from the inside of the abdomen and guides the hypodermic needle through the abdominal wall from the outside. When the needle point is visible through the peritoneum and almost enters the abdominal cavity, the surgeon retracts the needle around 5 mm. Then by deploying a test dose of the local anaesthetics a so called "Doyle's bulge" sign can confirm the right position in the nervous plane. A dose of 20 cc 3,75 mg/ml of Ropivacain is administered on each side of the abdominal wall in the midaxillary line, just in between the crista and costal margin.
  Interventions: Procedure: LAPTAP
- Ultrasound guided TAP block (Active Comparator): The anaesthesiologist uses ultrasound to identify the nervous plane in-between the external and transverse abdominal muscles. A dose of 20 cc 3,75 mg/ml of Ropivacain is administered on each side of the abdominal wall in the midaxillary line, just in between the crista and costal margin.
  Interventions: Procedure: LAPTAP

INTERVENTIONS:
Procedure: LAPTAP — Laparoscopic guided Transverse Abdominus Plane block

SUMMARY:
A randomized clinical trial aiming to compare two different techniques of performing a nerve blockage of the abdominal wall. When performing surgery on the colon and rectum surgeons often use a minimal invasive technique called Laparoscopic surgery. In this technique small incisions in the abdominal wall are used to put special ports trough into the abdomen so that surgical instrument can be inserted. To minimize the pain caused by these port-holes, a so-called Transversus Abdominus Plane (TAP) nerve block is performed directly after the surgery before the patient wakes up from narcosis.

This procedure is normally performed by the anesthesiologist using ultrasound to guide a needle to the right depth or "plane" in the abdominal wall where the nerves are gathered. When in the right position a local anesthetic is injected that will block the nerves and thereby anaesthetizing the abdominal wall for the first post-operative day.

Recently an alternative way of guiding the needle to the right position has been presented. By using a laparoscopic camera the surgeon can easily guide the needle and inject the local anesthetics during surgery. This way of performing the TAP block may save valuable time compared to the more cumbersome ultrasound guided technique while also not needing an extra anesthesiologist in the operating theater.

In this study we aim to include participants selected for elective minimal invasive surgery of the colon or rectum, where a TAP block is normally performed. The participant will be randomized to either a TAP block performed by the surgeon using laparoscopic guidance or by an anesthesiologist using ultrasound guidance. The intended surgery in itself will not be altered.

During surgery we will measure TAP procedure time, total surgical time, total duration of anesthesia and total time spent in the operating theater. The following 2 postoperative days we will measure experienced pain using a validated pain-score (VAS) and measure the total consumption of pain medication. 2 days after surgery the study ends for the participant and there is no further follow up.

By conducting this study we can determine whether a laparoscopic guided TAP by the surgeon, compared to a traditional ultrasound guided by the anesthesiologist; gives a shorter procedure time, shorter time of narcosis and reduced consumption of pain medications post-operative while still not affecting the experienced pain by the participant.

DETAILED DESCRIPTION:
At Danderyds hospital in Stockholm, since 2010, we are conducting patient care according to international evidence based Enhanced Recovery After Surgery (ERAS) protocols. Within colorectal surgery Danderyds hospital has been appointed ERAS Centre of Excellence due to documented favorable clinical results and a particularly suitable infrastructure for clinical research. The protocol comprises of 24 evidence-based interventions aimed at reducing so called surgical stress and promote early recovery after surgery. All interventions are executed in the same way for all patients. Optimal post-operative pain relief constitutes one of the 24 interventions and within this section a few methods are recommended. Transversus abdominus plane (TAP) block is one of those, and have been shown to reduce post-operative pain, reduce opioid consumption and elevate mobilization after surgery.

A TAP block is performed by injecting local anesthetics into the nervous plane in between the transverse and external muscles in the abdominal wall, and thereby blocking the nerves responsible for transmitting pain from the laparoscopic holes created during surgery.

Normally this TAP blockage is performed by the anesthesiologist using ultrasound to guide the needle for injection into the right plane of the abdominal wall. A procedure that can be cumbersome and that in our hospital setting takes around 30 minutes and is executed directly after the surgery but before the patient is alleviated of narcosis.

A novel technique has recently been described to guide the needle into the right position for the TAP block. In this technique the surgeon will use the laparoscopic camera and the port holes already made during surgery to visualize the inside of the abdominal wall, and by landmarks and a specially described bulging of the peritoneum as a marker, guide the needle from the outside and inject local anesthetics into the right plane. This method described by earlier studies has a procedure time at around 5+-1 minutes and has the benefit of not needing ultrasound or any other equipment not already present for the surgical procedure.

In this study we aim to include participants selected for elective robotic-assisted or laparoscopic minimal invasive surgery of the colon or rectum, where a TAP block is normally performed. The participant will be randomized to either a TAP block performed by the surgeon using laparoscopic guidance or by an anesthesiologist using ultrasound guidance. The intended surgery in itself will not be altered.

During surgery we will measure TAP procedure time, total surgical time, total duration of anesthesia and total time spent in the operating theater.

The following 2 postoperative days we will measure experienced pain using Visual Analog Scale (VAS) and measure the total opioid consumption. 2 days after surgery the study ends for the participant and there is no further follow up.

Previous studies on this technique have shown comparable or even better pain relieving efficacy compared to the ultrasound guided technique.

By conducting this study we can determine whether a laparoscopic guided TAP by the surgeon, compared to a traditional ultrasound guided TAP by the anesthesiologist; gives a shorter procedure time, shorter time of narcosis and reduced consumption of pain medications post-operative while still not affecting the experienced pain by the participant

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic or robot-assisted colorectal surgery.

Exclusion Criteria:

* IBD
* documented alcohol addiction
* documented opioid addiction
* unable to be assessed by Visual Analog Scale (cognitive impairment or other)
* Allergy against the local anaesthetic used, Ropivacain.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Post operative consumption of pain medication | 72 hours post surgery
  Difference in pain medication consumption between arms.
Visual Analog Scale | 72 hours post surgery
  Difference in experienced post operative pain using Visual Analog Scale (VAS) between arms. The VAS pain scale reaches from 0-10 where 0 equals No pain and 10 equals maximum pain.

SECONDARY OUTCOMES:
TAP procedure time | TAP procedure during surgery
  Time from start to finish of the TAP block between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Klas Pekkari, PhD, MD, Study Director — Danderyds Hospital, Karolinska Institute
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Laws in Sweden prohibits this.

REFERENCES:
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366
- [Background] Keller DS, Madhoun N, Ponte-Moreno OI, Ibarra S, Haas EM. Transversus abdominis plane blocks: pilot of feasibility and the learning curve. J Surg Res. 2016 Jul;204(1):101-8. doi: 10.1016/j.jss.2016.04.012. Epub 2016 Apr 27. PMID 27451874
- [Background] Keller DS, Ermlich BO, Schiltz N, Champagne BJ, Reynolds HL Jr, Stein SL, Delaney CP. The effect of transversus abdominis plane blocks on postoperative pain in laparoscopic colorectal surgery: a prospective, randomized, double-blind trial. Dis Colon Rectum. 2014 Nov;57(11):1290-7. doi: 10.1097/DCR.0000000000000211. PMID 25285696
- [Background] Favuzza J, Brady K, Delaney CP. Transversus abdominis plane blocks and enhanced recovery pathways: making the 23-h hospital stay a realistic goal after laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2481-6. doi: 10.1007/s00464-012-2761-y. Epub 2013 Jan 26. PMID 23355160
- [Background] Keller DS, Ermlich BO, Delaney CP. Demonstrating the benefits of transversus abdominis plane blocks on patient outcomes in laparoscopic colorectal surgery: review of 200 consecutive cases. J Am Coll Surg. 2014 Dec;219(6):1143-8. doi: 10.1016/j.jamcollsurg.2014.08.011. Epub 2014 Sep 16. PMID 25442068
- [Background] Tikuisis R, Miliauskas P, Lukoseviciene V, Samalavicius N, Dulskas A, Zabuliene L, Zabulis V, Urboniene J. Transversus abdominis plane block for postoperative pain relief after hand-assisted laparoscopic colon surgery: a randomized, placebo-controlled clinical trial. Tech Coloproctol. 2016 Dec;20(12):835-844. doi: 10.1007/s10151-016-1550-3. Epub 2016 Nov 28. PMID 27896461
- [Background] Walter CJ, Maxwell-Armstrong C, Pinkney TD, Conaghan PJ, Bedforth N, Gornall CB, Acheson AG. A randomised controlled trial of the efficacy of ultrasound-guided transversus abdominis plane (TAP) block in laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2366-72. doi: 10.1007/s00464-013-2791-0. Epub 2013 Feb 7. PMID 23389068
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Ravichandran NT, Sistla SC, Kundra P, Ali SM, Dhanapal B, Galidevara I. Laparoscopic-assisted Tranversus Abdominis Plane (TAP) Block Versus Ultrasonography-guided Transversus Abdominis Plane Block in Postlaparoscopic Cholecystectomy Pain Relief: Randomized Controlled Trial. Surg Laparosc Endosc Percutan Tech. 2017 Aug;27(4):228-232. doi: 10.1097/SLE.0000000000000405. PMID 28472015
- [Background] Zaghiyan KN, Mendelson BJ, Eng MR, Ovsepyan G, Mirocha JM, Fleshner P. Randomized Clinical Trial Comparing Laparoscopic Versus Ultrasound-Guided Transversus Abdominis Plane Block in Minimally Invasive Colorectal Surgery. Dis Colon Rectum. 2019 Feb;62(2):203-210. doi: 10.1097/DCR.0000000000001292. PMID 30540660
- [Background] Wong DJ, Curran T, Poylin VY, Cataldo TE. Surgeon-delivered laparoscopic transversus abdominis plane blocks are non-inferior to anesthesia-delivered ultrasound-guided transversus abdominis plane blocks: a blinded, randomized non-inferiority trial. Surg Endosc. 2020 Jul;34(7):3011-3019. doi: 10.1007/s00464-019-07097-y. Epub 2019 Sep 4. PMID 31485929
- [Background] Magee C, Clarke C, Lewis A. Laparoscopic TAP block for laparoscopic cholecystectomy: Description of a novel technique. Surgeon. 2011 Dec;9(6):352-3. doi: 10.1016/j.surge.2010.11.027. Epub 2010 Dec 24. No abstract available. PMID 22041649